CLINICAL TRIAL: NCT02705092
Title: Immediate Effect of Subliminal Priming With Subliminal Reward Stimuli on Standing Balance in Healthy Young Adults: A Randomized Controlled Trial
Brief Title: Immediate Effect of Subliminal Priming With Subliminal Reward Stimuli on Standing Balance in Healthy Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kibi International University (Other)
Responsible Party: Principal Investigator, Kazuki Hirao, PhD, OT, Assistant Professor, Kibi International University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 15-54
Record Dates: First submitted 2016-03-02; First posted 2016-03-10 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-06

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subliminal priming with subliminal reward stimuli (Experimental): This intervention consisted of five presentations [three cycles of mosaic (displayed for 117 ms each), physical exertion words as subliminal priming (displayed for 17 ms), and positive words as subliminal reward (displayed for 17 ms)].
  These were set to 1 package. 1 package is 24 times per 5 seconds presented in the animation (Animation of Skateboarding) for approximately 2 min.
  Interventions: Other: Subliminal priming with subliminal reward stimuli
- Subliminal priming with supraliminal reward stimuli (Experimental): This intervention consisted of four presentations [two cycles of mosaic (displayed for 117 ms each), physical exertion words as subliminal prime (displayed for 17 ms), and positive words as supraliminal reward (displayed for 150 ms)].
  These were set to 1 package. 1 package is 24 times per 5 seconds presented in the animation (Animation of Skateboarding) for approximately 2 min.
  Interventions: Other: Subliminal priming with supraliminal reward stimuli

INTERVENTIONS:
Other: Subliminal priming with subliminal reward stimuli — Positive words as subliminal reward (displayed for 17 ms).
  Arms: Subliminal priming with subliminal reward stimuli
Other: Subliminal priming with supraliminal reward stimuli — Positive words as supraliminal reward (displayed for 150 ms).
  Arms: Subliminal priming with supraliminal reward stimuli

SUMMARY:
The purpose of the study was to examine the immediate effect of subliminal priming with subliminal reward stimuli on standing balance in healthy young adults. The study also compared the outcomes with the immediate effects of subliminal priming with supraliminal reward stimuli.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers between 18 and 24 years of age
2. Males and Females

Exclusion Criteria:

1. Physical impairment, hindering performance of daily activities

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in the dynamic standing balance | Baseline and immediately after the intervention protocol
  Dynamic standing balance as measured by the Functional Reach Test

SECONDARY OUTCOMES:
Change in the static standing balance | Baseline and immediately after the intervention protocol
  Static standing balance as measured by the One-leg standing time with the eyes closed (maximum of 120 seconds)

CONTACTS AND LOCATIONS:
Overall Officials: Kazuki Hirao, PhD, OT, Principal Investigator — Kibi International University

IPD SHARING:
Plan to Share IPD: No